CLINICAL TRIAL: NCT07272070
Title: The Effect of Home-Based Walking on Symptoms and Health Profile of Hemodialysis Patients:Randomized Controlled Trial
Brief Title: The Effect of Home-Based Walking on Symptoms and Health Profile of Hemodialysis Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Figen Akay (Other)
Responsible Party: Sponsor-Investigator, Figen Akay, Specialist Nurse, Eskisehir Osmangazi University
Organization: Eskisehir Osmangazi University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: TABED 2-25-942
Record Dates: First submitted 2025-11-18; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Muscle Cramp; Hemodialysis; Vibration; Stretching
MeSH Terms: conditions — Muscle Cramp

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Home-based walking) (Experimental): Home-based walking
  Interventions: Other: Group A (Home-based walking)
- Group B (Usual hemodialysis care ) (Experimental): Usual hemodialysis care
  Interventions: Other: Group B (Usual hemodialysis care )

INTERVENTIONS:
Other: Group A (Home-based walking) — Verbal and written consent was obtained from patients who met the sampling criteria. At the first meeting, the Dialysis Symptom Index and Nottingham Health Profile will be assessed. Information was given about the pedometer tracking form and things to consider for walking exercises at home. Patients were asked to choose comfortable, lightweight athletic shoes that would hug their feet. The patient will be asked to walk on flat ground at home and wear cotton, non-sweaty clothes. It is necessary to walk forward at a moderate intensity 5 days a week. It will be explained that 6,000 steps should be taken in the first week and increased by 10% the following week. During the hemodialysis session, the tracking form will be checked with the pedometer application on the patient's smartphone. This group of patients will be asked to answer again in the 1st and 2nd months to see the change in the Dialysis Symptom Index and Nottingham Health Profile.
  Arms: Group A (Home-based walking)
Other: Group B (Usual hemodialysis care ) — Before starting the study, verbal and written consent will be obtained from patients who meet the sampling criteria. Patient identification forms will be completed. At the initial visit, patients' Dialysis Symptom Index and Nottingham Health Profile will be assessed, and this assessment will be recorded as week 0. Patients will be instructed to record their step count on the pedometer section of their smartphone at the end of each day. During each hemodialysis session, researchers will check the follow-up form using the pedometer application on the patient's smartphone and discuss daily care practices. This group of patients will be asked to answer again in the 1st and 2nd months to see the change in the Dialysis Symptom Index and Nottingham Health Profile.
  Arms: Group B (Usual hemodialysis care )

SUMMARY:
This study aims to evaluate the effect of 8 weeks of home-based moderate-speed walking on hemodialysis symptoms and health profile while patients are receiving hemodialysis treatment.

Due to permanent deterioration in kidney function, patients need hemodialysis treatment, which is the most commonly used treatment method among renal replacement therapies. Hemodialysis treatment causes a series of physical and psychological problems. Problems such as hypotension, headache, nausea, muscle cramps, itching and pain are physical problems, while depression, anxiety, cognitive disorders and stress are psychological problems. In addition, it has been reported that long-term hemodialysis treatment and all the resulting problems increase the tendency to a sedentary lifestyle in this patient group, leading to a decrease in physical function and activity, and indirectly to a low quality of life and low survival rates. For this reason, hemodialysis patients have difficulty meeting their daily activities and needs, and their dependency and healthcare burden increase. Adopting a sedentary lifestyle by these patients prevents them from managing both the physical and psychological problems of hemodialysis and their conditions such as hypertension and diabetes mellitus, and causes the disease to progress. Physical exercises, which are considered among the useful therapeutic suggestions in addition to pharmacological treatments in the management of the negative situations that arise, are considered as an easy, useful and effective intervention method. Kidney Disease: Improving Global Outcomes (KDIGO) recommends 30 minutes of moderate-intensity physical exercise at least 5 days a week. Additionally, it should not be overlooked that whether patients have places to do physical activity and what their facilities are are a detail that should be questioned by health professionals. Patients without suitable accommodations should be encouraged to engage in physical activity, especially in indoor spaces like home. Home-based walking exercise is known to be easy, inexpensive, and safe, and is also advantageous when the weather is not favorable. When we examined the studies in which home-based walking exercise was performed, it was determined that its effect on functional capacity was generally investigated, but its effect on the health outcomes and symptoms of patients receiving hemodialysis treatment was not evaluated. There was no evidence that home-based walking exercise had any effect on symptoms in patients receiving HD treatment. Therefore, it was planned to conduct a study to evaluate whether home-based walking exercise has an effect on patient health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients who agreed to participate in the research during the data collection process,
* Over 18 years of age,
* Speak and understand Turkish,
* Are at least literate,
* Can perform daily living activities independently,
* Own a smartphone.

Exclusion Criteria:

* Do not have sufficient cognitive ability,
* Have arthritic or orthopedic problems requiring assistance with walking,
* Have significant visual or hearing impairments,
* Walk regularly,
* Have a hemoglobin level <8 mg/dl,
* Have Stage IV of New York heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Dialysis symptoms | From enrollment to the end of treatment at 8 weeks
  The presence of dialysis symptoms is answered with a "yes" or "no" response. The scores obtained are summed to determine the scale score. The minimum score on this scale is "0" and the maximum is "150."
Health profile | From enrollment to the end of treatment at 8 weeks
  The Nottingham Health Profile consists of two sections. The first section covers the individual's health domain, and the second section covers areas affected by their health status. Questions are answered with "yes" or "no." The minimum score on the scale is "0," indicating good health, and the maximum score is "100," indicating poor health.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Machfer A, Fekih N, Ammar A, Hassen HBH, Daab W, Amor HH, Bouzid MA, Chtourou H. Effects of neuromuscular electrical stimulation during hemodialysis on muscle strength, functional capacity and postural balance in patients with end-stage renal disease: a randomized controlled trial. BMC Nephrol. 2025 Feb 19;26(1):86. doi: 10.1186/s12882-025-03994-8. PMID 39972246
- [Result] Manfredini F, Mallamaci F, D'Arrigo G, Baggetta R, Bolignano D, Torino C, Lamberti N, Bertoli S, Ciurlino D, Rocca-Rey L, Barilla A, Battaglia Y, Rapana RM, Zuccala A, Bonanno G, Fatuzzo P, Rapisarda F, Rastelli S, Fabrizi F, Messa P, De Paola L, Lombardi L, Cupisti A, Fuiano G, Lucisano G, Summaria C, Felisatti M, Pozzato E, Malagoni AM, Castellino P, Aucella F, Abd ElHafeez S, Provenzano PF, Tripepi G, Catizone L, Zoccali C. Exercise in Patients on Dialysis: A Multicenter, Randomized Clinical Trial. J Am Soc Nephrol. 2017 Apr;28(4):1259-1268. doi: 10.1681/ASN.2016030378. Epub 2016 Dec 1. PMID 27909047
- [Result] Koh KP, Fassett RG, Sharman JE, Coombes JS, Williams AD. Effect of intradialytic versus home-based aerobic exercise training on physical function and vascular parameters in hemodialysis patients: a randomized pilot study. Am J Kidney Dis. 2010 Jan;55(1):88-99. doi: 10.1053/j.ajkd.2009.09.025. Epub 2009 Nov 22. PMID 19932545
- [Result] Hiraki K, Shibagaki Y, Izawa KP, Hotta C, Wakamiya A, Sakurada T, Yasuda T, Kimura K. Effects of home-based exercise on pre-dialysis chronic kidney disease patients: a randomized pilot and feasibility trial. BMC Nephrol. 2017 Jun 17;18(1):198. doi: 10.1186/s12882-017-0613-7. PMID 28623895
- [Result] Fletcher BR, Damery S, Aiyegbusi OL, Anderson N, Calvert M, Cockwell P, Ferguson J, Horton M, Paap MCS, Sidey-Gibbons C, Slade A, Turner N, Kyte D. Symptom burden and health-related quality of life in chronic kidney disease: A global systematic review and meta-analysis. PLoS Med. 2022 Apr 6;19(4):e1003954. doi: 10.1371/journal.pmed.1003954. eCollection 2022 Apr. PMID 35385471